CLINICAL TRIAL: NCT03792204
Title: the Prevalence of "Wearing-off" in Patients With Parkinson's Disease in Shanghai, China: a Cross-sectional Investigation
Brief Title: the Prevalence of "Wearing-off" in Patients With Parkinson's Disease in Shanghai
Acronym: shapd-woq
Status: Completed | Type: Observational
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: XH-18-011
Record Dates: First submitted 2018-07-22; First posted 2019-01-03 (Actual); Last update posted 2019-01-03 (Actual); Status verified 2018-07

CONDITIONS: Wearing Off Effect; Parkinson Disease
Keywords: wearing off; wearing-off 9 questionnaire; prevalence; sensitivity; specificity
MeSH Terms: conditions — Parkinson Disease; Hypersensitivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD patients with wearing-off effect: people who have been clinically diagnosed with Parkinson's disease (PD) and have received anti PD therapy would be recruited into the study. The anti -PD treatment would not be changed in the population of the participants.
  We would use the tool of 'Wearing-off 9 questionnaire' to determine the prevalence of Wearing-off phenomenon in Parkinson's patients in Shanghai
  Interventions: Diagnostic Test: Wearing-off 9 questionnaire

INTERVENTIONS:
Diagnostic Test: Wearing-off 9 questionnaire — The participants would receive appropriate anti-PD medical treatments according to the patients' need during the investigation.The anti -PD treatment would not be changed in the population of the participants.
  Other Names: No other intervention

SUMMARY:
The study would be designed as a multi-center cross-sectional investigation on the prevalence of Wearing-off in Parkinson's patients in Shanghai as well as related influencing factors.

DETAILED DESCRIPTION:
PD patients would be randomly recruited into this investigation from around thirty hospital covering the 16 districts of Shanghai. The wearing off would be defined by two methods: the doctors' judgement or the WOQ-9 questionnaire which was a patient-determining tool. The investigation also includes the medicine, the severity of PD symptoms, the demographic factors. The study would be designed with the purpose of clarifying the prevalence of the "wearing-off" and its related influencing factors.

ELIGIBILITY:
Inclusion Criteria:

* have been clinical diagnosed with Parkinson's disease
* have received stable anti-Parkinson's treatment before being recruited to the study.

Exclusion Criteria:

* being suspicious of atypical Parkinson syndrome or secondary Parkinson syndromes
* have not received anti Parkinsonian treatment.
* being combined with serious cognitive dysfunction or psychiatric symptoms
* unable to complete the investigations.

Ages: 35 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: clinical diagnosed PD patients
Sampling Method: Probability Sample
Enrollment: 1480 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
the prevalence of wearing off effect in Parkinson's patients that received stable anti Parkinsonian therapy in Shanghai of China | 1 year
  every participant receives a clinical assessment of the wearing-off symptoms by a physician and completes a self rating scale of the wearing-off 9 questionnaire (WOQ-9) to obtain a prevalence of wearing-off positive individuals( wearing-off would be diagnosed by physicians during the clinical assessments)

SECONDARY OUTCOMES:
the sensitivity and the specificity of the wearing-off 9 questionnaire in the diagnosis of wearing-off effect in Parkinson's disease. | 1 year
  The physician assessment served as the standard for comparison with the WOQ-9 questionnaire. Sensitivity was defined as the probability that a PD patient, classified as having wearing-off (WO) according to physician assessment, would be classified as having the WO using the WOQ-9 questionnaire. The specificity was defined as the probability that a PD patient without the WO by physician assessments would be classified as being without the WO using the WOQ-9 questionnaire
the risk factors of wearing-off in Parkinson disease | 1 year
  assess patients clinical characteristics and medical treatments, including the onset age, disease duration and daily levodopa dosage in the subsets of Parkinson patients with wearing-off diagnosed by physician assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Liu, Ph.D., Study Chair — Xinhua hosipital affiliated to Shanghai Jiaotong university school of medicine
Locations (1):
- Xinhua hospital affiliated to Shanghai jiaotong university school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided to make individual participant data available to other researchers